CLINICAL TRIAL: NCT07303647
Title: Expression of Genes Related to Bone Metabolism in Saliva of Patients During Early Fixed Orthodontic Treatment: a Prospective Clinical Study
Brief Title: Genes Associated With Bone Metabolism in the Saliva During Orthodontic Treatment
Status: Active, not recruiting | Type: Observational
Sponsor: Kurdistan Higher Council of Medical Specialties (Other)
Responsible Party: Principal Investigator, Shehab Ahmed Hamad, professor, Kurdistan Higher Council of Medical Specialties
Other Study IDs: 2561
Record Dates: First submitted 2025-12-07; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Gene Expression Profiling; Orthodentic Appliances

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: PCR — Unstimulated whole saliva collection SOP (time of day, fasting, avoid toothbrushing immediately prior).
  RNA stabilization and extraction (saliva RNA kits).
  cDNA synthesis and quantitative RT-PCR (or RNA-seq if budget allows).
  Housekeeping genes for normalization (e.g., GAPDH, ACTB - validate stability in saliva).
  Analysis method: ΔΔCt → fold change.

SUMMARY:
Understanding the biological events during fixed orthodontic treatment is essential for optimizing treatment strategies, predicting patient response, and minimizing adverse effects. Most studies on bone remodeling have used invasive sampling methods such as tissue biopsies or serum collection; these methods cannot be used for routine clinical monitoring. Saliva is a simple medium that can reflect changes in local periodontal and bone conditions, it is also non-invasive and cheap. There is little evidence about the temporal expression of genes related to bone metabolism (RANKL, OPG, ALP, TRAP, RUNX2) in saliva during orthodontic therapy. This study will help advance the understanding of biological responses during orthodontic tooth movement and explore whether saliva can be an appropriate diagnostic medium for monitoring bone remodeling in orthodontic patients

ELIGIBILITY:
Inclusion criteria:

1.15 to 25 years of age 2.moderate crowding (3-6 mm) 3.generally good health with no systemic conditions that could influence bone metabolism 4. no recent use of medications known to affect bone metabolism (such as bisphosphonates and corticosteroids) or any other NSAIDs.

Exclusion criteria:

1. periodontal disease
2. smoking or any form of tobacco use
3. pregnancy or lactation
4. prior orthodontic treatment
5. craniofacial syndromes
6. The use of antibiotics within 3 months before the study. -

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Twenty-four patients (mean age 18.5 ± 3.2 years) who were receiving fixed orthodontic care were enrolled in this investigation.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2025-10-12 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
salivary genes of bone metabolism | 4 weeks
  Change in salivary gene expression levels of key bone-metabolism genes (e.g., RANKL, OPG, RUNX2, ALPL, BMP2) from baseline (T0) to subsequent timepoints during fixed orthodontic treatment, measured as ΔCt or fold-change (ΔΔCt) using qRT-PCR.

CONTACTS AND LOCATIONS:
Locations (1):
- Hawler teaching hospital, Erbil, Ervil, Iraq

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nugraha AP, Ernawati DS, Narmada IB, Bramantoro T, Riawan W, Situmorang PC, Nam HY. RANK-RANKL-OPG expression after gingival mesenchymal stem cell hypoxia preconditioned application in an orthodontic tooth movement animal model. J Oral Biol Craniofac Res. 2023 Nov-Dec;13(6):781-790. doi: 10.1016/j.jobcr.2023.10.009. Epub 2023 Nov 8. PMID 38028229